CLINICAL TRIAL: NCT00329667
Title: An Observational, Prospective Evaluation of the SJM Epic Valve
Brief Title: Observational Study of Prosthetic Tissue Aortic and Mitral Heart Valve
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sr. Director, Clinical, St. Jude Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSD 0206
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Valvular Heart Disease
Keywords: heart valve; mitral; aortic; valvular disease
MeSH Terms: conditions — Heart Valve Diseases

INTERVENTIONS:
Device: EPIC — Surgical replacement of a diseased, damaged, or malfunctioning native or prosthetic aortic and/or mitral heart valves

SUMMARY:
This study is a multi-center, prospective, non-randomized, observational study. The objectives of this study are to confirm the clinical safety and efficacy of the SJM Epic valve.

DETAILED DESCRIPTION:
This study is a multi-centered, multi-country, prospective, non-randomized, observational study, without concurrent or matched controls, conducted under a common protocol. Bayesian methods will be used for the design and analysis of this study. The Bayesian model will determine if the data for the valve configurations are poolable. Bayesian methods also provide a means of determining the appropriate stopping time for the study based on the amount of information generated. The objectives of this study are to confirm the clinical safety and efficacy of the SJM Epic Valve by establishing the following:

* adverse effect rates
* clinical status as indicated by NYHA functional classification
* hemodynamic performance

ELIGIBILITY:
Inclusion Criteria:

* The patient requires replacement of the aortic and/or mitral valve (Note: Patients undergoing concomitant procedures, e.g. coronary artery bypass grafting, valve repair, are eligible for this study).
* The patient (or legal guardian) has signed a study-specific informed consent, agreeing to the data collection and follow-up requirements.
* The patient is of legal age in host country.

Exclusion Criteria:

* Patient already has a prosthetic valve, other than the aortic and/or mitral valve being replaced at this time.
* The patient requires replacement of the tricuspid or pulmonary valve.
* The patient is pregnant or nursing.
* Patient has active endocarditis.
* Patient is actively participating in the study of an investigational drug or device.
* Patient has had an acute preoperative neurological event.
* The patient is undergoing renal dialysis.
* Patient is an intravenous drug abuser, alcohol abuser or prison inmate.
* Patient has an inability or unwillingness to return for the required follow-up intervals.
* The patient had the SJM Epic Valve implanted during the clinical study but then had the bioprosthesis explanted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2003-01; Primary Completion 2006-03 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Adverse effect rates | Ongoing
Clinical status as indicated by NYHA functional classification | At required follow-up visits
Hemodynamic performance | At required follow-up visits